CLINICAL TRIAL: NCT06925659
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of QLM2011 in Patients With Advanced Solid Tumors
Brief Title: A Study of QLM2011 in Subjects With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical (Hainan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QLM2011-101
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLM2011 (Experimental)
  Interventions: Drug: QLM2011
- Taxotere® (Experimental)
  Interventions: Drug: Taxotere®

INTERVENTIONS:
Drug: QLM2011 — QLM2011l by intravenous infusion.
  Arms: QLM2011
Drug: Taxotere® — Taxotere® by intravenous infusion
  Arms: Taxotere®

SUMMARY:
This trial is an open-label, single-center, dose-escalation and cohort-expansion Phase I clinical study in patients with advanced solid tumors. The purposeaim of this study is designed to evaluate the safety, tolerability, pharmacokinetics and preliminary antitumor activity of QLM2011 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18, ≤80 years, no gender limitation；
* Histologically or cytologically confirmed diagnosis of advanced or metastatic solid tumors, for which standard therapy either does not exist or has proven to be ineffective, intolerable for the patient；
* At least one measurable lesion as per RECIST version 1.1；
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1；
* Life expectancy ≥3 months；
* All subjects of reproductive potential must agree to use an effective method of contraception during the study and for 3 months after the last dose, and women of reproductive age must have a negative blood pregnancy result within 7 days prior to the first dose.

Exclusion Criteria:

* Chemotherapy, radiotherapy, targeted therapy， endocrine therapy, immunotherapy and other anti-tumor treatment within 28 days of the first dose of the study drug, 6 weeks for nitrosoureas or mitomycin C, 2 weeks (or 5 half-lives whichever is longer) for using fluorouracil or small molecule targeted drugs, 2 weeks for using traditional Chinese medicine with anti-tumor indications.
* Uncontrolled or clinically symptomatic serous cavity effusions (e.g., pericardial effusion, pleural effusion, ascites, etc.) requiring repeated puncture drainage or medical intervention.
* Toxicity from prior antitumor therapy has not recovered to ≤ Grade 1 per the Common Terminology Criteria for Adverse Events (CTCAE v5.0) (exceptions include alopecia, peripheral neuropathy, isolated laboratory abnormalities, or other toxicities deemed by the investigator to pose no safety risk).
* Have a history of other malignant tumors within 3 years before signing the informed consent, excluding cervical carcinoma in situ, basal cell carcinoma of the skin, papillary thyroid carcinoma or squamous cell carcinoma of the skin that has received radical treatment;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 21 days
  The DLT of QLM2011 will be determined.
Maximum tolerated dose (MTD) | up to 1 years
  The maximum tolerated dose (MTD) (if available) of QLM2011.
recommended Phase 2 dose (RP2D) | up to 1 years
  recommended Phase 2 dose (RP2D) of QLM2011.